CLINICAL TRIAL: NCT02423278
Title: The Long-term Effect of D4 Lymphadenectomy for Gastric Cancer: a Multicenter, Open-label, Randomized Trial
Brief Title: The Long-term Effect of D4 Lymphadenectomy for Gastric Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yulong He, Director of Center of Gastrointestinal Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010006
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Gastric Cancer; Surgery; Effects of Chemotherapy
Keywords: gastrectomy; lymphadenectomy; gastric cancer; adjuvant chemotherapy; overall survival
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D4 Lymphadenectomy (Experimental): This is the interventional group in which additional para-aortic lymph nodes are dissected meanwhile.
  Under this arm, main therapeutic measures are listed as follows:
  * three-cycle SOX chemo regimen (S-1+Oxaliplatin) as neoadjuvant chemotherapy
  * radical gastrectomy plus D4 lymphadenectomy
  * five-cycle SOX chemo as adjuvant chemotherapy
  * five-year follow-up program to evaluate the prognosis.
  Interventions: Procedure: Radical Gastrectomy Plus D4 Lymphadenectomy; Drug: S-1+Oxaliplatin
- D2 Lymphadenectomy (Experimental): This is the control group in which a classic surgical procedure for gastric cancer is performed.
  Under this arm, main therapeutic measures are included as follows:
  * three-cycle SOX chemo regimen (S-1+Oxaliplatin) as neoadjuvant chemotherapy
  * radical gastrectomy plus D2 lymphadenectomy (Without para-aortic lymph nodes dissection)
  * five-cycle SOX chemo as adjuvant chemotherapy
  * five-year follow-up program to evaluate the prognosis.
  Interventions: Procedure: Radical Gastrectomy Plus D2 Lymphadenectomy; Drug: S-1+Oxaliplatin

INTERVENTIONS:
Procedure: Radical Gastrectomy Plus D2 Lymphadenectomy — This surgical procedure is performed by the same high-experienced surgical team as the control arm.
  All lymph nodes around stomach (station 1&2 LNs) must be removed to achieve a radical lymphadenectomy. Para-aortic lymph nodes should not be dissected even if a suspected lymph node metastasis is diagnosed from radiographic exams.
  Other Names: D2 Lymphadenectomy
  Arms: D2 Lymphadenectomy
Procedure: Radical Gastrectomy Plus D4 Lymphadenectomy — This surgical procedure is also performed by the same high-experienced surgical team as the control arm.
  Lymph nodes around stomach (station 1&2 LNs) and para-aortic lymph nodes must be removed during the operation.
  Other Names: D4 Lymphadenectomy
  Arms: D4 Lymphadenectomy
Drug: S-1+Oxaliplatin — A perioperative chemotherapy, known as SOX regimen, should be performed in each enrolled patient with three-cycle treatments followed after a pathological carcinoma diagnosis. After a radical operation (arm groups), additional five-cycle treatments of adjuvant chemotherapy (SOX regimen) would be performed, followed by follow-up program. The treatment bundles are listed as follows:
  * S-1: 40~60mg bid，po, Day1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid）
  * Oxaliplatin: 130mg/m2，iv drip for 2h，Day1
  Other Names: SOX chemo Regimen

SUMMARY:
The main purpose of this study is to evaluate the effect of extensive lymphadenectomy procedure in treatment of gastric cancer. This study is designed as a open-label, multi-centers, randomized controlled trial. The overall survival and free disease survival are primary outcomes, with postoperative complication, hospital charges, and life quality as secondary outcomes.

DETAILED DESCRIPTION:
Background: Gastric cancer is the second leading cause of cancer-associated death worldwide, with high incidence in China. The prognosis of advanced gastric cancer is quite poor. Although perioperative chemotherapy may help to prolong survival in cases of advanced disease, radical tumor resection remains the most effective treatment for curable gastric cancer. Nowadays, radical gastrectomy with extended (D2) lymphadenectomy has become the standard for treatment of advanced gastric cancer. However, this surgical procedure cannot achieve a radical tumor resection for most cases with advanced disease. Hence, a more extensive (D2 plus para-aortic nodal dissection, D4) lymphadenectomy along with gastrectomy has been performed in Japan and other Asian countries. A recent study by Sasako et al. indicated that a prophylactic D4 lymphadenectomy did not improve the prognosis of curable gastric cancer, but increased the blood loss and operation time compared with single D2 procedure. We reviewed our database, which had collected almost 2,000 gastric cancer cases since its establishment in 1994, and found that the D4 surgical procedure actually improved the prognosis of T4 tumor and tumor with lymph node metastasis at the second stations. To further confirm the results from our retrospective analysis, we performed a prospective study with multicenter, open-label, and randomized design in the affiliated hospitals of Sun Yat-sen University. This study would be helpful to improve the prognosis of patients with advanced gastric cancer, and find more efficient management for curable gastric cancer.

Method: This study, which started from January, 2011 and planned to close after ten years, has been approved by the ethic committee of Sun Yat-sen University, with written inform consent obtained from all enrolled subjects. Patients who had histologically proven gastric adenocarcinoma and confirmed lymph node metastasis to para-aortic nodes (<3 enlarged lymph nodes) were prospectively enrolled in this trial. A standard D2 lymphadenectomy or D4 procedure was randomly decided by a formal randomization program. The primary end point of this study was overall survival, defined as the time from randomization to death. The secondary end points were recurrence-free survival, postoperative complications, length of stay, and hospital charges. Recurrence-free survival was defined as the time from randomization to the first recurrence of cancer or death from any cause. The follow-up period would last for at least five years after the definitive operation.

Significance: This study would further confirm the efficacy of D2 plus para-aortic nodal dissection(PAND) procedure for management of advanced gastric cancer as compared with the classic D2 lymphadenectomy operation. Moreover, the therapeutic measures employed in current study may guide the future treatment of advanced gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed pathological diagnosis of gastric cancer and visible para-aortic lymph nodes metastasis.
* Endurable D2/D4 gastrectomy and neoadjuvant chemotherapy.
* With moderate/good ECOG health rating (PS): 0-1 score.

Exclusion Criteria:

* Pregnant woman or lactating woman.
* With confirmed distant metastasis in liver, lung, bones, or other organs.
* Intolerable operation or neoadjuvant chemotherapy.
* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | five years after surgery
Relapse-free Survival | five years after surgery

SECONDARY OUTCOMES:
Early complications | within the first 30 days after surgery
  Rate of early postoperative events, such as anastomotic leak, intra-abdominal hemorrhage, adhesive intestinal obstruction and surgical site infection, in each arm.
Perioperative mortality | within the first 30 days after surgery
Life quality measured by HRQOL score | five years after surgery
  a questionnaire form would be sent to each enrolled patients after surgery.
Length of Hospital stay | an expected average of 4 weeks after admission
  The duration between admission and final discharge from hospital. An average of 4 weeks is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Yulong He, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China